CLINICAL TRIAL: NCT06173310
Title: DCE-MRI Guided Neoadjuvant Chemotherapy for Borderline Resectable Pancreatic Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Harrison Kim, Professor, Division of Advanced Medical Imaging Research, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 300012110
Record Dates: First submitted 2023-12-07; First posted 2023-12-15 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Borderline-resectable Pancreatic Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- borderline-resectable pancreatic cancer (BRPC) (Experimental)
  Interventions: Device: Point-of-care Portable Perfusion Phantom (P4)

INTERVENTIONS:
Device: Point-of-care Portable Perfusion Phantom (P4) — P4 is a perfusion phantom developed by Dr. Harrison Kim that can significantly reduce variation in quantitating perfusion of human abdominal tissues across MRI scanners.

SUMMARY:
The goal of this study is to test whether chemotherapy guided by a new imaging method named DCE-MRI can more effectively reduce a pancreatic tumor, enabling curable surgery, over the conventional method when a tumor is categorized as borderline resectable pancreatic cancer. UAB radiological research team has been studying a cutting-edge imaging technique named dynamic contrast-enhanced magnetic resonance imaging, or DCE-MRI, for over 10 years. This technique has been globally used to calculate the blood flow of various tissues, including tumors. Blood flow often serves as a critical indicator showing a disease status. For example, a pancreatic tumor typically has low blood flow, so it can be used as an indicator to identify the presence of a pancreatic tumor. In addition, an effective therapy can result in the increase of blood flow in a pancreatic tumor during the early period of treatment. Therefore, the investigators may be able to determine whether the undergoing therapy is effective or not by measuring the change of blood flow in the pancreatic tumor and deciding whether to continue the therapy or try a different one.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age 19 years or older).
* Patients with newly diagnosed and untreated borderline resectable pancreatic cancer.
* Patients with signed informed consent.

Exclusion Criteria:

* Any history of prior radiation or chemotherapy or surgical removal for pancreatic cancer.
* Participants with safety contraindications to MRI examination (determined by standard clinical screening).
* Participants who are pregnant, lactating or are planning to become pregnant during the study.
* Participants who are planning to father a child during the study.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-10-10 (Actual); Primary Completion 2029-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
To measure the reproducibility of qDCE-MRI measurement of BRPC. | 6 weeks +/- 2 weeks
  The pharmacokinetic (PK) parameter within the region of interest (ROI) will be averaged at each scan after P4-based error correction, and the mean values of two scans will be compared to calculate the reproducibility coefficient (%RDC) using the equation, %RDC=2.77wCV, where wCV is the within-subject coefficient of variation. The %RDC before P4-based error correction will also be calculated for comparison. Data reproducibility will be assessed using the intra-class correlation coefficient (ICC) as well. ICC = σ 2b / (σ 2b+ σ 2w), where σb is between-subject standard deviation and σw is within-subject standard deviation.

CONTACTS AND LOCATIONS:
Overall Officials: Harrison Kim, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (2):
- United States (2):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Indiana University Medical Center, Indianapolis, Indiana

IPD SHARING:
Plan to Share IPD: No